CLINICAL TRIAL: NCT02626065
Title: Immune Modulation Study in Patients With Metastatic Melanoma Treated With Anti-PD1 Monoclonal Antibodies
Acronym: PAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014.884
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Anti-PD1 monoclonal antibodies; Immune modulation; BRAF
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nivolumab, patients with BRAF mutation (Experimental): Nivolumab (dose equal to 3mg/kg), 10 mg/ml solution for infusion. injection of Nivolumab every two weeks from day 0 and until relapse, toxicity motivating withdrawal or temporary suspension of treatment or up to 54 weeks.
  Blood sampling at different time
  Interventions: Biological: blood sampling; Drug: Nivolumab
- Nivolumab, patients with BRAF wild type (Experimental): Nivolumab (dose equal to 3mg/kg), 10 mg/ml solution for infusion. injection of Nivolumab every two weeks from day 0 and until relapse, toxicity motivating withdrawal or temporary suspension of treatment or up to 54 weeks.
  Blood sampling at different time
  Interventions: Biological: blood sampling; Drug: Nivolumab

INTERVENTIONS:
Biological: blood sampling — Blood samples (44mL) will be taken before starting treatment with Nivolumab and at week 2, week 12, week 54 or at relapse (before week 54)
Drug: Nivolumab — injection of Nivolumab every two weeks from day 0 and until relapse, toxicity motivating withdrawal or temporary suspension of treatment or up to 54 weeks.

SUMMARY:
This is an open mono-centric prospective non-randomized study in patients with metastatic melanoma treated with Anti-PD1 monoclonal antibodies (Nivolumab). The aim of the study is to identify the immune cells modulations differences between patients who present a complete, partial or stable response and patients who have non-response to the therapy in order to establish an improving response rate strategy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years
* Patient with metastatic or unresectable melanoma
* Anti-PD1 monoclonal antibodies treatment indication
* Patient affiliated to a social security regime
* Signed Written Informed Consent.
* agree with the storage of his biological samples
* Women of childbearing potential must as mentioned in the summary of product characteristics (SPC) using two effective methods of contraception during treatment, and men whose partner is of childbearing potential must use effective contraception during treatment. For all patients treated men and women, contraception should be continued during the four months following the discontinuation of nivolumab.

Exclusion Criteria:

* development of haematological tumor during treatment
* Patients requiring concomitant chronic treatment with systemic corticosteroids or other immunosuppressive agents
* Patients with autoimmune disease.
* Patient with Occular melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
change the absolute number of dendritic cells before treatment and on treatment | before treatment (week 0), at week 2, at week 12, at week 54 or at relapse (before 54 weeks)
  absolute number / mm 3 of dendritic cells
change the percentage of cells producing cytokines in dendritic cells before treatment and on treatment | before treatment (week 0), at week 2, at week 12, at week 54 or at relapse (before 54 weeks)
  % of cells producing cytokines in dendritic cells
change the absolute number of subpopulations of T lymphocytes before treatment and on treatment | before treatment (week 0), at week 2, at week 12, at week 54 or at relapse (before 54 weeks)
  absolute number / mm 3 of different subpopulations of T lymphocyte
change the absolute number of monocytes before treatment and on treatment | before treatment (week 0), at week 2, at week 12, at week 54 or at relapse (before 54 weeks)
  absolute number / mm 3 of monocytes
change the percentage of cells producing cytokines in subpopulations of T lymphocytes before treatment and on treatment | before treatment (week 0), at week 2, at week 12, at week 54 or at relapse (before 54 weeks)
  % of cells producing cytokines in subpopulations of T lymphocytes
change the percentage of cells producing cytokines in monocytes before treatment and on treatment | before treatment (week 0), at week 2, at week 12, at week 54 or at relapse (before 54 weeks)
  % of cells producing cytokines in monocytes

SECONDARY OUTCOMES:
correlation between biological parameters and progression-free survival | progression between the date of first injection of immunotherapy and week 54 based on RECIST and ir-RECIST criterion
  absolute number / mm 3 of different population of cells and % of cells producing cytokines in the different population of cells will be correlated with the progression free survival
correlation between biological parameters on overall survival | death between the date of first injection of immunotherapy and week 54
  absolute number / mm 3 of different population of cells and % of cells producing cytokines in the different population of cells will be correlated with the overall survival
Identify predictive factors of overall response rate at week 12 based on RECIST and ir-RECIST criteria | response evaluation at week 12
  predictive factors like histological and cytological initial tumor type, initial immunological status will be evaluated at inclusion and correlated with the response
impact of treatments received prior to inclusion in the study on the biological parameters before and on treatment | antitumor treatment received from diagnosis of melanoma to inclusion
  absolute number / mm 3 of different population of cells and % of cells producing cytokines in the different population of cells will be correlated with treatments received prior to inclusion
correlation between the occurrence of autoimmune side effects and the biological parameters before and on treatment | occurence of autoimmune side effects from day 0 to week 54
  absolute number / mm 3 of different population of cells and % of cells producing cytokines in the different population of cells will be correlated with autoimmune side effects, based on CTCAE classification

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Background] Dalle S, Verronese E, N'Kodia A, Bardin C, Rodriguez C, Andrieu T, Eberhardt A, Chemin G, Hasan U, Le-Bouar M, Caramel J, Amini-Adle M, Bendriss-Vermare N, Dubois B, Caux C, Menetrier-Caux C. Modulation of blood T cell polyfunctionality and HVEM/BTLA expression are critical determinants of clinical outcome in anti-PD1-treated metastatic melanoma patients. Oncoimmunology. 2024 Jun 26;13(1):2372118. doi: 10.1080/2162402X.2024.2372118. eCollection 2024. PMID 38939518